CLINICAL TRIAL: NCT05358444
Title: Family Diabetes Prevention Program Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00310219; 1K23DK119581-01A1 (NIH)
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Results first posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: PreDiabetes; Overweight and Obesity; Type 2 Diabetes; Overweight, Childhood; Obesity, Childhood; Lifestyle, Healthy
Keywords: Prediabetes; Diabetes Prevention; Child obesity; Child overweight; Obesity; Overweight; Lifestyle Change
MeSH Terms: conditions — Prediabetic State; Overweight; Obesity; Diabetes Mellitus, Type 2; Pediatric Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes Prevention Program (DPP) (Active Comparator): Adult participants who are engaged in the Centers for Disease Control and Prevention's (CDC) National Diabetes Prevention Program lifestyle intervention (DPP) as delivered by the Johns Hopkins Brancati Center; this is a 12-month long, group-based lifestyle intervention, delivered by a certified lifestyle coach using a CDC-approved curriculum. This "concurrent control" group will consist of adults who are enrolled in the Brancati Center's DPP within 6 months of the intervention group start dates, who have children less than 18 years of age living in their households.
  Interventions: Behavioral: National Diabetes Prevention Program Lifestyle Intervention (DPP)
- Family Diabetes Prevention Program (Family DPP) (Experimental): Adult participants will engage in the family-oriented Diabetes Prevention Program lifestyle intervention (Family DPP); this is an augmented version of the DPP lifestyle intervention. This 12-month, group-based lifestyle intervention will include all elements of the DPP lifestyle intervention as delivered by the Johns Hopkins Brancati Center using a CDC-approved curriculum, with additional child-focused sessions in which adult participants will learn about children's health-related behaviors. Children will be present at the child-focused sessions and family activities, and will be engaged in data collection. These groups will be "mixed," in that non-study participants (adults who are eligible for the DPP), may also participate.
  Interventions: Behavioral: Family Diabetes Prevention Program (Family DPP)

INTERVENTIONS:
Behavioral: National Diabetes Prevention Program Lifestyle Intervention (DPP) — The National Diabetes Prevention Program lifestyle intervention (DPP) is a 12-month long, group-based lifestyle intervention for adults at high-risk for type 2 diabetes. The DPP will be delivered by certified coaches from the Johns Hopkins Brancati Center. The program uses the CDC's Prevent T2 curriculum, with a total of 32-34 sessions delivered over a 12-month period. In the initial "core" period (first 6 months), there are at least 16 sessions delivered on a weekly basis. In the "post-core" period, additional (at least 6) sessions are offered over a 6 month period. Sessions are delivered either in-person or via a virtual synchronous platform (Zoom).
  Arms: Diabetes Prevention Program (DPP)
Behavioral: Family Diabetes Prevention Program (Family DPP) — The Family DPP has been developed as an augmented version of the National Diabetes Prevention Program Lifestyle Intervention (DPP). It includes all elements of the 12-month, group-based DPP lifestyle intervention, led by a CDC certified-coach using a CDC-approved curriculum (involving around 32-34 sessions). The augmentations of the Family DPP supplement the DPP's sessions to additionally address barriers to adults' own lifestyle change efforts related to being a caregiver of children AND to introduce basic concepts regarding healthy child habits related to dietary intake, physical activity and screen time, and sleep. The Family DPP will involve thus additional sessions that will be delivered to the adult DPP participant, and in which children, ages 5 through 12, may also be engaged.
  Arms: Family Diabetes Prevention Program (Family DPP)

SUMMARY:
This study will examine the feasibility and acceptability of a family-oriented augmentation of the Diabetes Prevention Program lifestyle intervention (DPP), called the Family DPP. It will also preliminarily examine adult and child health and health behavior outcomes. The DPP is a 12-month, group-based lifestyle intervention for adults at high-risk for type 2 diabetes, in which adult participants learn skills and strategies to achieve the program's goals of 5% weight loss and 150 minutes/week of moderate-vigorous physical activity. The Family DPP will consist of all elements of the evidence-based DPP, along with augmentations including additional child-focused sessions in which adult participants will learn about principles and strategies for promoting healthy lifestyle behaviors in children, ages 5 through 12 years. Children may participate in certain child-focused sessions, too. The non-randomized pilot feasibility study will consists of 2 arms/groups: 1) the concurrent "control" group, consisting of adults who are enrolled in the DPP; and 2) the "intervention" arm, in which the adult participants will engage in the Family DPP (and children may participate in certain aspects of the Family DPP focused on children). The study will recruit 10-15 adult-child dyads, for the "intervention" groups, and 10-15 adults for the concurrent control group. In addition to data collected from adult participants as a routine part of the DPP, the study will examine additional adult health behaviors and health outcomes and child health outcomes (change in body mass index z-score) and health behaviors at baseline, 6 months and 12 months (program end) among participants in the "intervention" group.

ELIGIBILITY:
Inclusion Criteria for the Intervention Arm:

* For ADULT participants, inclusion criteria are:

  1. Meeting eligibility criteria for the CDC's National Diabetes Prevention Program lifestyle intervention, which are:

     1. 18 years of age and older;
     2. not pregnant at time of enrollment;
     3. body mass index (BMI) of ≥25 kg/m2 (≥23 kg/m2 , if of Asian race);
     4. meet one of the following: a) have prediabetes (defined as fasting glucose of 100-125 mg/dL; plasma glucose measured 2 hours after 75 gm glucose load of 140 to 199 mg/dL, or A1c of 5.7% to 6.4%); b) history of clinically diagnosed gestational diabetes mellitus (GDM) during a previous pregnancy; c) high risk for diabetes based on CDC or American Diabetes Association (ADA) Diabetes Screening Test).

     AND
  2. being a primary caregiver of at least one eligible child aged 5 through 12 years at time of recruitment (defined as caring for the child, with a responsibility for the child's food, sleep and activity habits, at least 3 days out of the week)
* For CHILD participants, inclusion criteria are:

  1. being aged 5 through 12 years at time of recruitment;
  2. not having a medical condition which leads to inability to comply with general pediatric dietary or physical activity goals; AND
  3. not concurrently enrolled in a structured weight management program.

Exclusion Criteria for Intervention Arm:

* For ADULT participants, exclusion criteria include

  1. Conditions that would exclude their participation in the DPP lifestyle intervention which include:

     1. pregnancy;
     2. having end-stage renal disease;
     3. having type 1 or type 2 diabetes.
  2. They will also be excluded if they are concurrently enrolled in a structured weight management program.
* For CHILD participants: exclusion criteria include:

  1. having a medical condition which leads to inability to comply with general pediatric dietary or physical activity goals;
  2. being enrolled in a structured weight management program.

     For the Control Arm/Concurrent Control Group, this will only enroll ADULT participants.
* The inclusion criteria are:

  1. Being a participant in the Brancati Center's Diabetes Prevention Program, in a group that has started within 6 months of Intervention Arm group start
  2. Lives with a child less than 18 years of age in their household

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maya S Venkataramani, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Background] Damschroder LJ, Moin T, Datta SK, Reardon CM, Steinle N, Weinreb J, Billington CJ, Maciejewski ML, Yancy WS Jr, Hughes M, Makki F, Richardson CR. Implementation and evaluation of the VA DPP clinical demonstration: protocol for a multi-site non-randomized hybrid effectiveness-implementation type III trial. Implement Sci. 2015 May 12;10:68. doi: 10.1186/s13012-015-0250-0. PMID 25962598
- [Background] Taveras EM, Mitchell K, Gortmaker SL. Parental confidence in making overweight-related behavior changes. Pediatrics. 2009 Jul;124(1):151-8. doi: 10.1542/peds.2008-2892. PMID 19564295
- [Background] Golan M. Fifteen years of the Family Eating and Activity Habits Questionnaire (FEAHQ): an update and review. Pediatr Obes. 2014 Apr;9(2):92-101. doi: 10.1111/j.2047-6310.2013.00144.x. Epub 2013 Feb 28. PMID 23447444

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study enrolled adult participants only in the DPP arm, and adult-child dyads in the Family DPP arm. 10 adult participants were enrolled in the DPP arm, and 12 adult-child dyads were enrolled in the Family DPP arm (12 adults and 12 children).
Groups:
- Family Diabetes Prevention Program (Family DPP): Adult participants will engage in the family-oriented Diabetes Prevention Program lifestyle intervention (Family DPP); this is an augmented version of the DPP lifestyle intervention. This 12-month, group-based lifestyle intervention will include all elements of the DPP lifestyle intervention as delivered by the Johns Hopkins Brancati Center using a CDC-approved curriculum, with additional child-focused sessions in which adult participants will learn about children's health-related behaviors. Children will be present at the child-focused sessions and family activities, and will be engaged in data collection. Groups will be "mixed," in that non-study participants (adults who are eligible for the DPP), may also participate.
  Family DPP: The Family DPP has been developed as an augmented version of the National Diabetes Prevention Program Lifestyle Intervention (DPP). It includes all elements of the 12-month, group-based DPP lifestyle intervention, led by a CDC certified-coach using a CDC-approved curriculum (involving around 32-34 sessions). The augmentations of the Family DPP include 2 additional sessions that address barriers to adults' own lifestyle change efforts related to being a caregiver of children and child-focused sessions to introduce basic concepts regarding healthy child lifestyle habits. The additional sessions that will be delivered to the adult DPP participant, and in which children, ages 5 through 12, can also be engaged.
Period: Overall Study
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Started | 10 (10 Adult participants) | 12 (12 adult-child dyads (dyad= 1 adult and 1 child per dyad))
Completed (Completion defined as completing the 12 month study data collection point) | 10 (10 Adult participants) | 8 (8 adult-child dyads (dyad= 1 adult and 1 child per dyad))
Not Completed | 0 | 4
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Population: This study enrolled adult participants only in the DPP arm, and adult-child dyads in the Family DPP arm. 10 adult participants were enrolled in the DPP arm, and 12 adult-child dyads were enrolled in the Family DPP arm (12 adults and 12 children, for a total of 24 participants in the Family DPP arm).
Groups:
- Total: Total of all reporting groups
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP) | Total
Number analyzed (Participants) | 10 | 24 | 34
Age, Categorical [Count of Participants; unit: Participants] — Population: Adult participants only were enrolled in the DPP arm. Child participants and adult participants (as adult-child dyads) were enrolled in the Family DPP arm.
  Participants
    Adult participants: number analyzed (Participants) | 10 | 12 | 22
    Adult participants: <=18 years | 0 | 0 | 0
    Adult participants: Between 18 and 65 years | 9 | 11 | 20
    Adult participants: >=65 years | 1 | 1 | 2
    Child participants: number analyzed (Participants) | 0 | 12 | 12
    Child participants: <=18 years |  | 12 | 12
    Child participants: Between 18 and 65 years |  | 0 | 0
    Child participants: >=65 years |  | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] — Population: Adult participants only were enrolled in the DPP arm. Child participants and adult participants (as adult-child dyads) were enrolled in the Family DPP arm.
  years
    Adult participants: number analyzed (Participants) | 10 | 12 | 22
    Adult participants | 48.2 [37 to 71] | 46.4 [34 to 70] | 47.2 [34 to 71]
    Child participants: number analyzed (Participants) | 0 | 12 | 12
    Child participants |  | 9.85 [5.40 to 12.81] | 9.85 [5.4 to 12.81]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Adult participants only were enrolled in the DPP arm. Child participants and adult participants (as adult-child dyads) were enrolled in the Family DPP arm.
  Participants
    Adult participants: number analyzed (Participants) | 10 | 12 | 22
    Adult participants: Female | 8 | 10 | 18
    Adult participants: Male | 2 | 2 | 4
    Child participants: number analyzed (Participants) | 0 | 12 | 12
    Child participants: Female |  | 9 | 9
    Child participants: Male |  | 3 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Adult participants only were enrolled in the DPP arm. Child participants and adult participants (as adult-child dyads) were enrolled in the Family DPP arm.
  Participants
    Adult participants: number analyzed (Participants) | 10 | 12 | 22
    Adult participants: Hispanic or Latino | 0 | 0 | 0
    Adult participants: Not Hispanic or Latino | 9 | 11 | 20
    Adult participants: Unknown or Not Reported | 1 | 1 | 2
    Child participants: number analyzed (Participants) | 0 | 12 | 12
    Child participants: Hispanic or Latino |  | 0 | 0
    Child participants: Not Hispanic or Latino |  | 8 | 8
    Child participants: Unknown or Not Reported |  | 4 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Adult participants only were enrolled in the DPP arm. Child participants and adult participants (as adult-child dyads) were enrolled in the Family DPP arm.
  Participants
    Adult participants: number analyzed (Participants) | 10 | 12 | 22
    Adult participants: American Indian or Alaska Native | 0 | 0 | 0
    Adult participants: Asian | 0 | 0 | 0
    Adult participants: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Adult participants: Black or African American | 7 | 9 | 16
    Adult participants: White | 2 | 3 | 5
    Adult participants: More than one race | 1 | 0 | 1
    Adult participants: Unknown or Not Reported | 0 | 0 | 0
    Child Participants: number analyzed (Participants) | 0 | 12 | 12
    Child Participants: American Indian or Alaska Native |  | 0 | 0
    Child Participants: Asian |  | 0 | 0
    Child Participants: Native Hawaiian or Other Pacific Islander |  | 0 | 0
    Child Participants: Black or African American |  | 6 | 6
    Child Participants: White |  | 2 | 2
    Child Participants: More than one race |  | 0 | 0
    Child Participants: Unknown or Not Reported |  | 4 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 24 | 34
Adult participant/caregiver relation to child [Count of Participants; unit: Participants] — Population: This is a characteristic unique to adult participants only.
  Participants
    number analyzed (Participants) | 10 | 12 | 22
    Parent | 9 | 10 | 19
    Grandparent | 1 | 2 | 3
Adult participant/caregiver employment status [Count of Participants; unit: Participants] — Population: This is a characteristic unique to adult participants only.
  Participants
    number analyzed (Participants) | 10 | 12 | 22
    Employed/Works Outside the Home | 8 | 9 | 17
    Not Employed | 2 | 3 | 5
Household annual income, category [Count of Participants; unit: Participants] — Population: This is a household level characteristic (1 household per adult in the control arm, 1 household per adult-child dyad in the intervention arm).
  Participants
    number analyzed (Participants) | 10 | 12 | 22
    Less than $10,000 | 0 | 1 | 1
    Between $10,001 and $20,000 | 0 | 0 | 0
    Between $20,001 and $40,000 | 1 | 1 | 2
    Between $40,001 and $60,000 | 0 | 1 | 1
    Between $60,001 and $70,000 | 1 | 0 | 1
    Above $70,001 | 8 | 9 | 17
    Decline to answer | 0 | 0 | 0
Household receipt of benefits in past year [Number; unit: household] — As reported by adult participants for their households. Some households received more than one type of benefit Population: This is a household level characteristic (1 household per adult in the control arm, 1 household per adult-child dyad in the intervention arm).
  household
    None: number analyzed (Participants) | 10 | 12 | 22
    None | 6 | 9 | 15
    Special Supplemental Nutrition Program for Women, Infants and Children: number analyzed (Participants) | 10 | 12 | 22
    Special Supplemental Nutrition Program for Women, Infants and Children | 0 | 1 | 1
    Supplemental Nutrition Assistance Program: number analyzed (Participants) | 10 | 12 | 22
    Supplemental Nutrition Assistance Program | 1 | 3 | 4
    Temporary Cash Assistance/TANF: number analyzed (Participants) | 10 | 12 | 22
    Temporary Cash Assistance/TANF | 0 | 1 | 1
    Temporary Disability Assistance: number analyzed (Participants) | 10 | 12 | 22
    Temporary Disability Assistance | 0 | 0 | 0
    Energy Assistance: number analyzed (Participants) | 10 | 12 | 22
    Energy Assistance | 0 | 0 | 0
    Medicaid: number analyzed (Participants) | 10 | 12 | 22
    Medicaid | 3 | 3 | 6
    Reduced cost or free school lunch: number analyzed (Participants) | 10 | 12 | 22
    Reduced cost or free school lunch | 3 | 2 | 5
    Other: number analyzed (Participants) | 10 | 12 | 22
    Other | 1 | 1 | 2
    Decline to answer: number analyzed (Participants) | 10 | 12 | 22
    Decline to answer | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Adult Participant Attendance in Program as Assessed by Total Number of Required Program Sessions Attended, Core
Description: The average total number of required core period program sessions attended by the adult participant (inclusive of make-up sessions) including all DPP (and, if in Family DPP, additional Family DPP sessions); for Family DPP adult participants this will also be examined for the subset of DPP sessions and additional Family DPP sessions.
Time Frame: 6 months
Population: Adult participants in the DPP group and Family DPP group, who did not formally withdraw from the study.
Measure: Mean (Standard Error); unit: sessions
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 10 | 11
sessions
  All Core Sessions | 17.6 (0.22) | 14.8 (1.8)
  DPP only core sessions: number analyzed (Participants) | 0 | 11
  DPP only core sessions |  | 13.5 (1.6)
  Family DPP child-focused sessions: number analyzed (Participants) | 0 | 11
  Family DPP child-focused sessions |  | 1.4 (0.24)

2. Primary Outcome: Adult Participant Attendance in Program as Assessed by Total Number of Program Sessions Attended, Full Program
Description: The average total number of all required sessions attended by the adult participant (inclusive of make-up sessions); for Family DPP adult participants this will also be examined for the subset of DPP sessions only, and additional required Family DPP sessions only (of which there were 10), and didactic/required child-focused sessions only (of which there were 8).
Time Frame: 12 months
Population: Adult participants in the DPP group and Family DPP group, who did not formally withdraw from the study.
Measure: Mean (Standard Error); unit: sessions
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 10 | 11
sessions
  All required sessions | 25.2 (0.99) | 25.1 (3.9)
  All required DPP sessions: number analyzed (Participants) | 0 | 11
  All required DPP sessions |  | 18.8 (2.8)
  All required Family DPP sessions: number analyzed (Participants) | 0 | 11
  All required Family DPP sessions |  | 6.3 (1.2)
  All required child-focused Family DPP sessions: number analyzed (Participants) | 0 | 11
  All required child-focused Family DPP sessions |  | 4.9 (1.0)

3. Primary Outcome: Adult Participant Attendance in Program as Assessed by Percentage of Program Sessions Attended, Core
Description: The average percentage of required core period program sessions attended by the adult participant (inclusive of make-up sessions) in each arm (denomiator of 18 for DPP, and 20 for Family DPP); for Family DPP adult participants this will also be examined for the subset of required DPP sessions only (denominator is 18) and additional Family DPP sessions only (of which there were 2).
Time Frame: 6 months
Population: Adult participants in the DPP group and Family DPP group, who did not formally withdraw from the study.
Measure: Mean (95% Confidence Interval); unit: percentage of sessions
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 10 | 11
percentage of sessions
  Percentage of all required core sessions | 97.8 [95.0 to 100.0] | 74.1 [53.6 to 94.6]
  Percentage of all required core DPP sessions: number analyzed (Participants) | 0 | 11
  Percentage of all required core DPP sessions |  | 74.7 [54.5 to 95.0]
  Percentage of required core Family DPP sessions: number analyzed (Participants) | 0 | 11
  Percentage of required core Family DPP sessions |  | 68.2 [41.0 to 95.4]

4. Primary Outcome: Adult Participant Attendance in Program as Assessed by Percentage of Program Sessions Attended, Full Program
Description: The percentage of all required program sessions attended by the adult participant (inclusive of make-up sessions); for Family DPP adult participants this will also be examined for the subset of DPP sessions only, all additional Family DPP sessions only (of which there were 10), and child-focused DPP sessions only (of which there were 8).
Time Frame: 12 months
Population: Adult participants in the DPP group and Family DPP group, who did not formally withdraw from the study.
Measure: Mean (95% Confidence Interval); unit: percentage of sessions
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 10 | 11
percentage of sessions
  Percentage of all required sessions | 87.8 [80.2 to 95.4] | 64.3 [42.1 to 86.6]
  Percentage of all required DPP sessions: number analyzed (Participants) | 0 | 11
  Percentage of all required DPP sessions |  | 64.8 [43.4 to 86.4]
  Percentage of all required FDPP sessions: number analyzed (Participants) | 0 | 11
  Percentage of all required FDPP sessions |  | 62.8 [35.2 to 90.3]
  Percentage of all child-focused required FDPP sessions: number analyzed (Participants) | 0 | 11
  Percentage of all child-focused required FDPP sessions |  | 61.4 [32.4 to 90.3]

5. Primary Outcome: Child Participant Attendance in Family Diabetes Prevention Program
Description: The percentage of required child-focused sessions (N=8) attended by the child participant will be examined for child participants in the Family DPP arm only.
Time Frame: 12 months
Population: Child participants (who were enrolled in the Family DPP only), who did not formally withdraw from the study
Measure: Mean (95% Confidence Interval); unit: percentage of child-focused sessions
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 0 | 11
percentage of child-focused sessions |  | 44.3 [20.5 to 68.2]

6. Primary Outcome: Feasibility of Measurement of Child-related Outcomes as Assessed by the Percentage of Total Child Participants for Whom Data Are Collected
Description: The percentage of total enrolled child participants (in the intervention arm) for whom BMI data and also child-health behavior data are collected will be examined for at baseline data collection point.
Time Frame: Baseline
Population: Enrolled child participants in the Family DPP arm.
Measure: Number; unit: percentage of children
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 0 | 12
percentage of children |  | 100

7. Primary Outcome: Feasibility of Measurement of Child-related Outcomes as Assessed by the Percentage of Total Child Participants for Whom Data Are Collected
Description: The percentage of total enrolled child participants (in the Family DPP interventionarm) for whom BMI data and also child-health behavior data are collected will be examined for the 6 month data point.
Time Frame: 6 months
Population: Enrolled child participants in the Family DPP Arm, who had not formally withdrawn from the study.
Measure: Number; unit: percentage of children
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 0 | 11
percentage of children |  | 81.2

8. Primary Outcome: Feasibility of Measurement of Child-related Outcomes as Assessed by the Percentage of Total Child Participants for Whom Data Are Collected
Description: The percentage of total enrolled child participants (in the Family DPP intervention arm) for whom BMI data and child-health behavior data are collected will be examined for the 12 month data point.
Time Frame: 12 months
Population: There are no child participants in the DPP arm.
Measure: Number; unit: percentage of children
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 0 | 11
percentage of children |  | 72.7

9. Primary Outcome: Satisfaction With Family Diabetes Prevention Program as Assessed by Study Team Designed Questionnaire
Description: Mean Likert-scale score (for most items, Likert scale on a range of 1 to 4; from strongly disagree (1) to strongly agree (4)), exploring satisfaction with Family DPP content and structure). Mean of participant choice is reported.
Time Frame: 12 months (end of intervention)
Population: Adult participants in the Family DPP (intervention arm) only who completed the FDPP satisfaction survey.
Measure: Mean (Standard Error); unit: score on Likert scale (range 1 to 4)
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 0 | 8
score on Likert scale (range 1 to 4)
  "I would recommend the Family DPP to others" |  | 3.88 (0.13)
  "I believe the Family DPP sessions were helpful in helping me address children's health behaviors" |  | 3.75 (0.16)
  "I believe the Family DPP sessions were helpful in helping me address my own health behaviors" |  | 3.75 (0.16)

10. Primary Outcome: Intervention Fidelity as Assessed by a Fidelity Checklist
Description: Using an adapted DPP fidelity checklist, this will examine fidelity of delivery of Family DPP specific sessions; percentage of content delivered by coach during session is reported.
Time Frame: Up to 12 months
Population: The units analyzed are FDPP sessions.
Measure: Number (95% Confidence Interval); unit: percentage of session content
Units Other Than Participants: Family DPP specific sessions
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 0 | 12
Number analyzed (Family DPP specific sessions) | 0 | 14
percentage of session content |  | 91.4 [86.9 to 95.8]

11. Primary Outcome: Total Cost of Program Delivery
Description: Cost of program delivery (including staffing, materials, wrap-around support) per participant (or for FDPP, per dyad). Calculated separately for DPP and Family DPP (intervention) arm.
  Total delivery cost of DPP incurred by the delivering center was used for DPP cost/participant- this is calculated as a total cost for a set number of cohorts/participants, divided by number of participants. There is a single value (no variation) for each category of cost that was used to calculate this number, and thus no measure of precision or dispersion can be calculated due to nature of calculating a total cost.
  For FDPP dyads, additional costs related to FDPP intervention and delivery were included in this calculation.
Time Frame: 12 months (end of intervention)
Measure: Number; unit: dollar cost per participant
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 10 | 12
dollar cost per participant | 1022.95 | 1288.97

12. Primary Outcome: Recruitment Rate as Assessed by the Rate of Enrollment Per Week
Description: Recruitment rate is calculated as the number of eligible participants (adult controls or adult-child dyad intervention arm) consenting and completing enrollment and participating in the trial, divided by period of recruitment (in weeks). This value is calculated separately for intervention arm and concurrent control group. The measure is calculated as # of participants recruited (total)/total number of weeks of recruitment. (For intervention arm, 12 adult-child dyads/22 weeks; for control arm adults: 10 adults/9.5 weeks).
Time Frame: During recruitment period up to 22 weeks
Measure: Number; unit: adults enrolled per week
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 10 | 12
adults enrolled per week | 1.05 | 0.55

13. Primary Outcome: Survey Administration Feasibility as Assessed by Mean Time for Administration of Surveys to Participants
Description: Mean time (minutes) for administration of baseline surveys to adult participant and child participant in the Family DPP (intervention) arm.
Time Frame: Baseline
Population: Data was not able to be collected, as measurement of time required for administration was unable to be assessed by study team member while simultaneously administering surveys.
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 0 | 0

14. Primary Outcome: Survey Administration Feasibility as Assessed by Mean Time for Administration of Surveys to Participants
Description: Mean time (minutes) for administration of surveys to adult participant and child participant at 6 month time point in the Family DPP (intervention) arm.
Time Frame: 6 months
Population: as for outcome 13
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 0 | 0

15. Primary Outcome: Survey Administration Feasibility as Assessed by Mean Time for Administration of Surveys to Participants
Description: Mean time (minutes) for administration of surveys to adult participant and child participant in the Family DPP (intervention) arm.
Time Frame: 12 months
Population: as for outcome 13
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Percentage Change in Adult Participant Weight (Kilograms)
Description: Percentage change in weight (kilograms) from baseline to end of program (Self-report from home weight may be used depending on program delivery modality). Calculated for adults who are considered "DPP completers" (requires having been in DPP at least 9 months and also attending at least 8 sessions in core period) per the DPP specific definition.
Time Frame: Baseline and 12 months (end of intervention)
Population: Adults who are considered "DPP completers" (requires having been in DPP at least 9 months and also attending at least 8 sessions in core period) as per the DPP specific definition.
Measure: Mean (Standard Deviation); unit: percentage change in weight (kilograms)
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 9 | 7
percentage change in weight (kilograms) | -8.19 (1.97) | -3.83 (3.18)

17. Secondary Outcome: Change in Child Body Mass Index (BMI) Z-score
Description: Change in Centers for Disease Control and Prevention's extended Body Mass Index (BMI) z-score at end of program (12 months) compared to baseline and 6 months, from BMI calculated from weight and height measurements during program in the Family DPP (intervention) arm. (Z-score of 0 indicates population mean value).
  Calculated for all children and among subgroup of children with overweight or obese weight status at baseline.
Time Frame: Baseline, 6 months and 12 months (end of intervention)
Population: Children in the Family DPP (intervention) arm only who did not formally withdraw from the study and for whom data was collected at relevant time points; there were no children enrolled in the DPP (control) arm.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 0 | 11
z-score
  Change in BMI extended Z-score of all child participants, baseline to 12 months: number analyzed (Participants) | 0 | 8
  Change in BMI extended Z-score of all child participants, baseline to 12 months |  | 0.02 (0.31)
  Change in BMI extended Z-score of all child participants, 6 months to 12 months: number analyzed (Participants) | 0 | 8
  Change in BMI extended Z-score of all child participants, 6 months to 12 months |  | -0.017 (0.25)
  Change in BMI extended Z-score of child participants with overweight /obesity, baseline to 12 months: number analyzed (Participants) | 0 | 5
  Change in BMI extended Z-score of child participants with overweight /obesity, baseline to 12 months |  | 0.06 (0.32)
  Change in BMI extended Z-score of child participants with overweight /obesity, 6 months to 12 months: number analyzed (Participants) | 0 | 5
  Change in BMI extended Z-score of child participants with overweight /obesity, 6 months to 12 months |  | -0.019 (0.18)

18. Secondary Outcome: Adult Participant Physical Activity as Assessed by Average Duration of Activity Per Week
Description: Average number of minutes/week of moderate-vigorous physical activity by self report, at baseline.
Time Frame: Baseline
Population: This outcome was assessed among adult study participants in either the control or intervention arm for whom data was collected at the baseline time point AND who did not formally withdraw from the study.
Measure: Mean (Standard Deviation); unit: minutes of physical activity, per week
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 10 | 11
minutes of physical activity, per week | 147.4 (139.8) | 106.82 (126.22)

19. Secondary Outcome: Adult Participant Physical Activity as Assessed by Average Duration of Activity Per Week
Description: Average number of minutes/week of moderate-vigorous physical activity by self report, at 6 months (during core period) among adults for whom data was collected through this time point (this reflects average of values reported Sessions 2 through 18).
Time Frame: 6 months
Population: Among adult study participants for whom data was collected through the time point as described (and who did not formally withdraw from the study)
Measure: Mean (Standard Deviation); unit: minutes of physical activity per week
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 10 | 8
minutes of physical activity per week | 192.72 (110.27) | 137.11 (92.41)

20. Secondary Outcome: Adult Participant Physical Activity as Assessed by Average Duration of Activity Per Week
Description: Average number of minutes/week of moderate-vigorous physical activity by self report, by 12 months/end of program, among adults considered DPP completers (this reflects average of values reported Sessions 2 through 29).
Time Frame: 12 months
Population: Among adult study participants considered as per specific Diabetes Prevention Program definition to have been completers in the DPP.
Measure: Mean (Standard Deviation); unit: minutes of physical activity per week
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 9 | 7
minutes of physical activity per week | 188.97 (99.69) | 113.78 (67.38)

21. Secondary Outcome: Percentage of Adult Participants Who Met Physical Activity Achievement
Description: Whether or not the adult participant met the program goal of an average 150 minutes/week of moderate-vigorous physical activity.
Time Frame: 12 months
Population: Adult participants considered DPP completers.
Measure: Number; unit: percentage of participants
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 9 | 7
percentage of participants | 55.6 | 14.29

22. Secondary Outcome: Change in Adult Participant Dietary Pattern Related to Fruit and Vegetable Intake Frequency
Description: Questions from the Behavioral Risk Factor Surveillance System (BRFSS) 2017 modules on fruit, vegetable and fruit juice intake as assessed by participant recall (for 1 week period), which quantify frequency of intake of these food items over 1 week-recall period; changes in intake patterns from baseline, at 6 and 12 months, will be assessed for adults in the Family DPP (intervention) arm.
Time Frame: Baseline, 6 months and 12 months (end of intervention)
Population: This outcome was assessed among adult study participants in the intervention arm only; outcome was calculated for adult participants for whom data was collected at referenced time points (e.g., baseline and 6 months, and baseline and 12 months) AND who did not formally withdraw from the study.
  (This data was not collected in the control arm).
Measure: Mean (Standard Deviation); unit: number of times per day, in prior week
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 0 | 9
number of times per day, in prior week
  Change in Frequency of Total Fruit Intake, baseline to 6 months |  | -0.38 (1.01)
  Change in Frequency of Total Fruit Intake, baseline to 12 months: number analyzed (Participants) | 0 | 8
  Change in Frequency of Total Fruit Intake, baseline to 12 months |  | 0.30 (1.23)
  Change in Frequency of Total Vegetable Intake, baseline to 6 months |  | -.02 (0.87)
  Change in Frequency of Total Vegetable Intake, baseline to 12 months: number analyzed (Participants) | 0 | 8
  Change in Frequency of Total Vegetable Intake, baseline to 12 months |  | 0.02 (0.77)

23. Secondary Outcome: Change in Adult Participant Dietary Pattern Related to Sugary Beverage Intake Frequency
Description: Questions from the BRFSS on sugary beverage intake, as assessed by participant recall (for 1 week period), which quantify frequency of intake of sugary beverages over 1 week-recall period; changes in intake patterns from baseline, at 6 and 12 months, will be assessed for adults in the Family DPP (intervention) arm.
Time Frame: Baseline, 6 months and 12 months (end of intervention)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: number of times per day, in prior week
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 0 | 9
number of times per day, in prior week
  Change in Frequency of Sugary Beverage intake, baseline to 6 months |  | -0.10 (0.61)
  Change in Frequency of Sugary Beverage intake, baseline to 12 months |  | -0.07 (0.53)

24. Secondary Outcome: Change in Child Participant Fruit and Vegetable Intake Frequency
Description: Questions from the YRBS 2017 modules on fruit and vegetable intake, which quantify intake of these food items over a 7-day period; questions will be asked of caregivers of all child participants and directly of children ages 9 through 12 years. Changes in intake patterns from baseline will be assessed.
Time Frame: Baseline, 6 months and 12 months (end of intervention)
Population: This outcome was assessed among child study participants (in the intervention arm only; there were no children enrolled in the DPP (control arm); outcome was calculated for child participants for whom data was collected at referenced time points (e.g., baseline and 6 months, and baseline and 12 months) AND who did not formally withdraw from the study.
Measure: Mean (Standard Deviation); unit: number of times per day, in prior week
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 0 | 11
number of times per day, in prior week
  Change in Frequency of Total Fruit Intake, baseline to 6 months: number analyzed (Participants) | 0 | 9
  Change in Frequency of Total Fruit Intake, baseline to 6 months |  | 0.02 (1.95)
  Change in Frequency of Total Fruit Intake, baseline to 12 months: number analyzed (Participants) | 0 | 8
  Change in Frequency of Total Fruit Intake, baseline to 12 months |  | -0.68 (1.17)
  Change in Frequency of Total Fruit Intake, 6 months to 12 months: number analyzed (Participants) | 0 | 8
  Change in Frequency of Total Fruit Intake, 6 months to 12 months |  | -0.38 (1.79)
  Change in Frequency of Total Vegetable Intake, baseline to 6 months: number analyzed (Participants) | 0 | 9
  Change in Frequency of Total Vegetable Intake, baseline to 6 months |  | -0.57 (1.39)
  Change in Frequency of Total Vegetable Intake, baseline to 12 months: number analyzed (Participants) | 0 | 8
  Change in Frequency of Total Vegetable Intake, baseline to 12 months |  | -0.73 (1.51)
  Change in Frequency of Total Vegetable Intake, 6 months to 12 months: number analyzed (Participants) | 0 | 8
  Change in Frequency of Total Vegetable Intake, 6 months to 12 months |  | -0.21 (0.70)

25. Secondary Outcome: Change in Child Participant Sugary Beverage Intake Frequency
Description: Questions from the Youth Risk Behavioral Surveillance System (YRBSS) on sugary beverage intake frequency over a 7-day period; questions will be asked of caregivers of all child participants and directly of children ages 9 through 12 years. Changes in intake patterns from baseline, at 6 and 12 months, will be assessed.
Time Frame: Baseline, 6 and 12 months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: number of times per day, in prior week
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 0 | 11
number of times per day, in prior week
  Change in Frequency of Sugary Beverage Intake, baseline to 6 months: number analyzed (Participants) | 0 | 9
  Change in Frequency of Sugary Beverage Intake, baseline to 6 months |  | -0.08 (0.86)
  Change in Frequency of Sugary Beverage Intake, baseline to 12 months: number analyzed (Participants) | 0 | 8
  Change in Frequency of Sugary Beverage Intake, baseline to 12 months |  | -0.25 (1.39)
  Change in Frequency of Sugary Beverage Intake, 6 months to 12 months: number analyzed (Participants) | 0 | 8
  Change in Frequency of Sugary Beverage Intake, 6 months to 12 months |  | -0.21 (1.13)

26. Secondary Outcome: Change in Child Participant Screen Time
Description: Adaptation of questions from YRBSS regarding average number of hours of screen time/day, asked weekday or weekend over past 7 days. Questions will be asked of caregivers of all child participants and directly of children ages 9 through 12 years. (Options given of less than 1 hour, coded as 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours and 5 hours or more (coded as 5 hours). Changes in number of hours of screen time from baseline, at 6 and 12 months, will be assessed for children in the Family DPP (intervention) arm.
Time Frame: Baseline, 6 months and 12 months (end of intervention)
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: hours of screen time/day, over past week
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 0 | 11
hours of screen time/day, over past week
  Change in hours of sleep per night weekdays, baseline to 6 months: number analyzed (Participants) | 0 | 9
  Change in hours of sleep per night weekdays, baseline to 6 months |  | -0.28 (0.97)
  Change in hours of sleep per night weekdays, baseline to 12 months: number analyzed (Participants) | 0 | 8
  Change in hours of sleep per night weekdays, baseline to 12 months |  | -0.06 (0.56)
  Change in hours of sleep per night weekdays, 6 months to 12 months: number analyzed (Participants) | 0 | 8
  Change in hours of sleep per night weekdays, 6 months to 12 months |  | 0.13 (0.83)
  Change in hours of sleep per night weekends, baseline to 6 months: number analyzed (Participants) | 0 | 9
  Change in hours of sleep per night weekends, baseline to 6 months |  | -0.44 (0.88)
  Change in hours of sleep per night weekends, baseline to 12 months: number analyzed (Participants) | 0 | 8
  Change in hours of sleep per night weekends, baseline to 12 months |  | -0.25 (0.89)
  Change in hours of sleep per night weekends,6 months to 12 months: number analyzed (Participants) | 0 | 8
  Change in hours of sleep per night weekends,6 months to 12 months |  | 0.25 (0.89)

27. Secondary Outcome: Change in Child Participant Sleep Patterns
Description: Adaptation of questions from YRBSS regarding average number of hours of sleep per night on weekdays, over last week. Questions will be asked of caregivers of all child participants and directly of children ages 9 through 12 years. Changes will be assessed, at 6 and 12 months.
Time Frame: Baseline, 6 months and 12 months (end of intervention)
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: hours of sleep on weekday, past week
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 0 | 11
hours of sleep on weekday, past week
  Change in number of hours of sleep on weekday in past week, baseline to 6 months: number analyzed (Participants) | 0 | 9
  Change in number of hours of sleep on weekday in past week, baseline to 6 months |  | -0.83 (1.41)
  Change in number of hours of sleep on weekday in past week, baseline to 12 months: number analyzed (Participants) | 0 | 8
  Change in number of hours of sleep on weekday in past week, baseline to 12 months |  | -0.75 (1.39)
  Change in number of hours of sleep on weekday in past week, 6 months to 12 months: number analyzed (Participants) | 0 | 8
  Change in number of hours of sleep on weekday in past week, 6 months to 12 months |  | 0.25 (1.46)

28. Secondary Outcome: Change in Adult Caregiver Perceived Self-efficacy for Behavioral Change
Description: Questionnaire exploring confidence in achieving behavioral goals related to physical activity, sleep and dietary modifications, using a Likert scale with options from 1 to 5, higher scores indicating higher perceived self-efficacy). Mean change in self-efficacy for each item from baseline (to 6 months and 12 months) will be assessed for adults in the Family DPP (intervention) arm.
Time Frame: Baseline, 6 months and 12 months (end of intervention)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 0 | 11
score on a scale
  Change from baseline in self-efficacy to achieve 150 min mod-vigorous physical activity/week,at 6mo |  | 0.22 (1.20)
  Change from baseline in self-efficacy to achieve150 min mod-vigorous physical activity/week,at 12mo: number analyzed (Participants) | 0 | 8
  Change from baseline in self-efficacy to achieve150 min mod-vigorous physical activity/week,at 12mo |  | 0.37 (0.92)
  Change from baseline in self-efficacy for taking 2-min fitness break every 30 min when seated,at 6mo |  | 0 (1.22)
  Change from baseline in self-efficacy for taking 2-min fitness break every 30 min when seated,at 12m: number analyzed (Participants) | 0 | 8
  Change from baseline in self-efficacy for taking 2-min fitness break every 30 min when seated,at 12m |  | -0.25 (1.58)
  Change from baseline in self-efficacy for reducing sugary beverage intake, at 6mo |  | -0.33 (0.5)
  Change from baseline in self-efficacy for reducing sugary beverage intake, at 12mo: number analyzed (Participants) | 0 | 8
  Change from baseline in self-efficacy for reducing sugary beverage intake, at 12mo |  | -0.25 (0.46)
  Change from baseline in self-efficacy for getting 7 or more hours of sleep per night, at 6mo |  | 0 (1.66)
  Change from baseline in self-efficacy for getting more than 7 hours of sleep per night, at 12mo: number analyzed (Participants) | 0 | 8
  Change from baseline in self-efficacy for getting more than 7 hours of sleep per night, at 12mo |  | 0.75 (0.89)
  Change in self-efficacy for including non-starchy vegetable in meals daily, at 6mo |  | -0.22 (0.97)
  Change in self-efficacy for including non-starchy vegetable in meals daily, at 12mo |  | -0.125 (0.64)

29. Secondary Outcome: Change in Child Participant Physical Activity Levels
Description: Adaptations of questions from YRBS regarding number of days meeting physical activity goal/week. Questions will be asked of caregivers of all child participants and directly of children ages 9 through 12 years. Changes in activity patterns from baseline, including whether meeting daily physical activity guidelines, will be assessed for children in the Family DPP (intervention) arm.
Time Frame: Baseline, 6 months and 12 months (end of intervention)
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: number of days per week
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 0 | 11
number of days per week
  Change in number days/week achieving 60 minutes activity, over past week, baseline to 6 months |  | 0.11 (1.76)
  Change in number days/week achieving 60 minutes activity, over past week, baseline to 12 months |  | 0.88 (1.96)
  Change in number days/week achieving 60 minutes activity, over past week, 6 months to 12 months |  | 0.88 (2.53)

30. Secondary Outcome: Change in Parenting Self-efficacy for Child Health Behavior Change
Description: Questionnaire exploring adult caregiver confidence in supporting child to achieve behavioral goals related to physical activity, sleep, screen time and diet, using a Likert scale from 1 to 5 with higher scores indicating higher perceived self-efficacy). Mean change in parenting self-efficacy overall and for each item from baseline, at 6 and 12 months, will be assessed for adults in the Family DPP (intervention) arm.
Time Frame: Baseline, 6 months and 12 months (end of intervention)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: score on Likert scale (1-5)
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 0 | 11
score on Likert scale (1-5)
  Change from baseline in parenting self-efficacy for supporting child physical activity, at 6 mo |  | -0.33 (1)
  Change from baseline in parenting self-efficacy for supporting child physical activity, at 12mo: number analyzed (Participants) | 0 | 8
  Change from baseline in parenting self-efficacy for supporting child physical activity, at 12mo |  | 0.50 (1.07)
  Change from 6 mo in parenting self-efficacy for supporting child physical activity, at 12 mo: number analyzed (Participants) | 0 | 8
  Change from 6 mo in parenting self-efficacy for supporting child physical activity, at 12 mo |  | 1 (0.93)
  Change from baseline in parenting self-efficacy for limiting child screen time, at 6mo: number analyzed (Participants) | 0 | 8
  Change from baseline in parenting self-efficacy for limiting child screen time, at 6mo |  | -0.25 (0.71)
  Change from baseline in parenting self-efficacy for limiting child screen time, at 12mo: number analyzed (Participants) | 0 | 8
  Change from baseline in parenting self-efficacy for limiting child screen time, at 12mo |  | 0.38 (0.92)
  Change from 6mo in parenting self-efficacy for limiting child screen time, at 12mo: number analyzed (Participants) | 0 | 7
  Change from 6mo in parenting self-efficacy for limiting child screen time, at 12mo |  | 0.43 (0.54)
  Change from baseline in parenting self-efficacy for limiting child sugary beverage intake, at 6mo |  | -0.22 (1.20)
  Change from baseline in parenting self-efficacy for limiting child sugary beverage intake, at12 mo: number analyzed (Participants) | 0 | 8
  Change from baseline in parenting self-efficacy for limiting child sugary beverage intake, at12 mo |  | 0.25 (1.16)
  Change from 6mo in parenting self-efficacy for limiting child sugary beverage intake, at 12mo: number analyzed (Participants) | 0 | 8
  Change from 6mo in parenting self-efficacy for limiting child sugary beverage intake, at 12mo |  | 0.63 (1.06)
  Change from baseline in parenting self-efficacy for supporting child sleep, at 6mo: number analyzed (Participants) | 0 | 9
  Change from baseline in parenting self-efficacy for supporting child sleep, at 6mo |  | -0.67 (0.71)
  Change from baseline in parenting self-efficacy for supporting child sleep, at 12 mo: number analyzed (Participants) | 0 | 8
  Change from baseline in parenting self-efficacy for supporting child sleep, at 12 mo |  | 0 (0.93)
  Change from 6 mo in parenting self-efficacy for supporting child sleep, at 12mo: number analyzed (Participants) | 0 | 8
  Change from 6 mo in parenting self-efficacy for supporting child sleep, at 12mo |  | 0.63 (1.06)
  Change from baseline in parenting self-efficacy for supporting child fruit and veggie intake, at 6mo: number analyzed (Participants) | 0 | 9
  Change from baseline in parenting self-efficacy for supporting child fruit and veggie intake, at 6mo |  | 0 (0.87)
  Change from baseline in parenting self-efficacy for supporting child fruit and veggie intake,at 12mo: number analyzed (Participants) | 0 | 8
  Change from baseline in parenting self-efficacy for supporting child fruit and veggie intake,at 12mo |  | -0.13 (0.93)
  Change from 6mo in parenting self-efficacy for supporting child fruit and veggie intake, at 12mo: number analyzed (Participants) | 0 | 8
  Change from 6mo in parenting self-efficacy for supporting child fruit and veggie intake, at 12mo |  | -0.25 (0.89)

31. Secondary Outcome: Change in Family Eating/Activity Habits and Home Environment
Description: The Family Eating and Activity Habits Questionnaire-Revised (FEAHQ-R) is a 32-item, self-report instrument; score range 0-128 with likert scale options 0-4. It is a clinical tool that captures family member eating and activity habits and also factors related with obesity in the overall home environment for children and caregivers. A higher score is associated with less favorable or appropriate patterns. Mean changes in scores from baseline, at 6 and 12 months, will be assessed in the Family DPP (intervention) arm.
Time Frame: Baseline, 6 months and 12 months (end of intervention)
Population: This outcome was assessed among adult AND child study participants in the intervention arm only; outcome was calculated for adult and child participants for whom data was collected at referenced time points (e.g., baseline and 6 months, and baseline and 12 months) AND who did not formally withdraw from the study.
  (This data was not collected in the control arm).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 0 | 11
score on a scale
  Change from baseline in FEAHQ-R score for child, at 6 months: number analyzed (Participants) | 0 | 9
  Change from baseline in FEAHQ-R score for child, at 6 months |  | 3.33 (6.83)
  Change from baseline in FEAHQ-R score for child, at 12 months: number analyzed (Participants) | 0 | 8
  Change from baseline in FEAHQ-R score for child, at 12 months |  | 2.48 (10.07)
  Change from 6 months in FEAHQ-R score for child, at 12 months: number analyzed (Participants) | 0 | 8
  Change from 6 months in FEAHQ-R score for child, at 12 months |  | -1.40 (3.26)
  Change from baseline in FEAHQ-R score for adult, at 6 months |  | -1.86 (12.7)
  Change from baseline in FEAHQ-R score for adult, at 12 months |  | -7.38 (11.66)
  Change from 6 months in FEAHQ-R score for adult, at 12 months |  | -5.09 (11.29)

32. Secondary Outcome: Change in Caregiver Knowledge Regarding Child Health Behaviors
Description: Questionnaire examining knowledge or awareness of age-specific pediatric guidelines for sleep, dietary intake, screen time and physical activity. 4 total questions, with percentage of questions answered correctly ranging from 0% to 100%. Mean change in the percentage of questions answered correctly from baseline, will be examined for adults in the Family DPP (intervention) arm.
Time Frame: Baseline, 6 months and 12 months (end of intervention)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: percentage of questions answered correct
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 0 | 11
percentage of questions answered correct
  Change from baseline in percentage of questions answered correctly, at 6 months: number analyzed (Participants) | 0 | 9
  Change from baseline in percentage of questions answered correctly, at 6 months |  | 5.56 (30.0)
  Change from baseline in percentage of questions answered correctly, at 12 months: number analyzed (Participants) | 0 | 8
  Change from baseline in percentage of questions answered correctly, at 12 months |  | 25 (18.90)
  Change from 6 months in percentage of questions answered correctly, at 12 months: number analyzed (Participants) | 0 | 8
  Change from 6 months in percentage of questions answered correctly, at 12 months |  | 21.88 (33.91)

33. Secondary Outcome: Change in Caregiver Attitudes Regarding Child Health Behaviors
Description: Questionnaire examining caregiver beliefs and attitudes towards age-specific guidelines for sleep, dietary intake, screen time and physical activity, using a Likert scale for extent to which respondent agrees or disagrees with statements (Likert Scale Options of 1-4: 1-Strongly Disagree to 4-Strongly Agree). Higher score indicates higher agreement with the statement. Mean change in score for each from baseline examined for adults in the Family DPP (intervention) arm.
Time Frame: Baseline, 6 months and 12 months (end of intervention)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: change in Likert scale score
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
Number analyzed (Participants) | 0 | 11
change in Likert scale score
  Change from baseline in degree of agreement that child is at a healthy weight, at 6 months: number analyzed (Participants) | 0 | 8
  Change from baseline in degree of agreement that child is at a healthy weight, at 6 months |  | 0 (0.53)
  Change from baseline in degree of agreement that child is at a healthy weight, at 12 months: number analyzed (Participants) | 0 | 8
  Change from baseline in degree of agreement that child is at a healthy weight, at 12 months |  | 0.38 (0.52)
  Change from 6 months in degree of agreement that child is at a healthy weight, at 12 months: number analyzed (Participants) | 0 | 7
  Change from 6 months in degree of agreement that child is at a healthy weight, at 12 months |  | 0.29 (0.49)
  Change from baseline in degree of agreement that child gets enough sleep, at 6 months: number analyzed (Participants) | 0 | 8
  Change from baseline in degree of agreement that child gets enough sleep, at 6 months |  | -0.13 (0.35)
  Change from baseline in degree of agreement that child gets enough sleep, at 12 months: number analyzed (Participants) | 0 | 8
  Change from baseline in degree of agreement that child gets enough sleep, at 12 months |  | -0.25 (0.46)
  Change from 6 months in degree of agreement that child gets enough sleep, at 12 months: number analyzed (Participants) | 0 | 8
  Change from 6 months in degree of agreement that child gets enough sleep, at 12 months |  | -0.13 (0.35)
  Change from baseline in degree of agreement that child is as active as they need to be, at 6 months: number analyzed (Participants) | 0 | 9
  Change from baseline in degree of agreement that child is as active as they need to be, at 6 months |  | -0.22 (1.20)
  Change from baseline in degree of agreement that child is as active as they need to be, at 12 months: number analyzed (Participants) | 0 | 8
  Change from baseline in degree of agreement that child is as active as they need to be, at 12 months |  | 0.25 (1.04)
  Change from 6 months in degree of agreement that child is as active as they need to be, at 12 months: number analyzed (Participants) | 0 | 8
  Change from 6 months in degree of agreement that child is as active as they need to be, at 12 months |  | 0.25 (0.46)
  Change from baseline in degree of agreement that child eats enough fruits and veggies, at 6 months: number analyzed (Participants) | 0 | 9
  Change from baseline in degree of agreement that child eats enough fruits and veggies, at 6 months |  | 0.11 (0.60)
  Change from baseline in degree of agreement that child eats enough fruits and veggies, at 12 months: number analyzed (Participants) | 0 | 8
  Change from baseline in degree of agreement that child eats enough fruits and veggies, at 12 months |  | 0 (0.93)
  Change from 6 months in degree of agreement that child eats enough fruits and veggies, at 12 months: number analyzed (Participants) | 0 | 8
  Change from 6 months in degree of agreement that child eats enough fruits and veggies, at 12 months |  | -0.13 (1.13)
  Change from baseline in degree of agreement that child needs to cut down sugary bev, at 6 months: number analyzed (Participants) | 0 | 9
  Change from baseline in degree of agreement that child needs to cut down sugary bev, at 6 months |  | -0.78 (0.97)
  Change from baseline in degree of agreement that child needs to cut down sugary bev, at 12 months: number analyzed (Participants) | 0 | 8
  Change from baseline in degree of agreement that child needs to cut down sugary bev, at 12 months |  | -0.63 (1.19)
  Change from 6 months in degree of agreement that child needs to cut down sugary bev, at 12 months: number analyzed (Participants) | 0 | 8
  Change from 6 months in degree of agreement that child needs to cut down sugary bev, at 12 months |  | 0.13 (0.99)
  Change from baseline in degree of agreement that child needs to cut screen time, at 6 months: number analyzed (Participants) | 0 | 9
  Change from baseline in degree of agreement that child needs to cut screen time, at 6 months |  | -0.33 (0.87)
  Change from baseline in degree of agreement that child needs to cut screen time, at 12 months: number analyzed (Participants) | 0 | 8
  Change from baseline in degree of agreement that child needs to cut screen time, at 12 months |  | -0.63 (1.19)
  Change from 6 months in degree of agreement that child needs to cut screen time, at 12 months: number analyzed (Participants) | 0 | 8
  Change from 6 months in degree of agreement that child needs to cut screen time, at 12 months |  | -0.38 (0.52)
  Change from baseline in degree of agreement that child's weight puts at risk for diabetes, at 6 mo: number analyzed (Participants) | 0 | 9
  Change from baseline in degree of agreement that child's weight puts at risk for diabetes, at 6 mo |  | 0.56 (0.73)
  Change from baseline in degree of agreement that child's weight puts at risk for diabetes, at 12 mo: number analyzed (Participants) | 0 | 8
  Change from baseline in degree of agreement that child's weight puts at risk for diabetes, at 12 mo |  | 0.25 (0.46)
  Change from 6 months in degree of agreement that child's weight puts at risk for diabetes, at 6 mo: number analyzed (Participants) | 0 | 8
  Change from 6 months in degree of agreement that child's weight puts at risk for diabetes, at 6 mo |  | -0.38 (0.52)

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: Serious or Potentially Serious Adverse Events were defined as:
  1) Event that was life threatening, or placed the pt at immediate risk of death; 2) Event that caused persistent or significant disability/incapacity (lasted at least 1 month and changed the pt's life); 3) Event that required or prolonged a hospitalization; 4) Pregnancy that resulted in congenital anomaly or birth defect; 5) Death; 6) Event that caused other significant hazards/potentially serious harm to research subjects/others.
Arm/Group | Diabetes Prevention Program (DPP) | Family Diabetes Prevention Program (Family DPP)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/10 | 3/24
Other Adverse Events (participants affected / at risk) | 0/10 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diabetes Prevention Program (DPP) (N=10) | Family Diabetes Prevention Program (Family DPP) (N=24)
Musculoskeletal injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Fracture of ankle. Not related to intervention.
Hospitalization (Gastrointestinal disorders) | 1 (1) | 0 (0) — Not related to intervention.
Musculoskeletal injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Vertebral fracture. Not related to intervention.
Elective surgery (Surgical and medical procedures) | 0 (0) | 1 (1) — Not related to intervention.

LIMITATIONS AND CAVEATS:
The focus of this trial was to examine measures of feasibility and acceptability related to the Family DPP and delivery of the intervention. The overall small sample size does not allow for definitive measurement of impact on health behaviors and health outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT05358444/Prot_SAP_000.pdf